CLINICAL TRIAL: NCT05554146
Title: The Impact of Medical Cannabis on Pain and Inflammation in People Living With HIV
Brief Title: Pain Inflammation and Cannabis in HIV
Acronym: PITCH-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Colorado, Boulder (Other); University of Pittsburgh (Other); Vireo Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-13662; K23DA053997 (NIH)
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections; Neuropathic Pain; Cannabis
MeSH Terms: conditions — HIV Infections; Neuralgia; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: We will observe participants who are enrolled in one of 4 arms in a partnering study over 14 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Coupon for a Discounted Placebo Product (Other): We will observe participants who were previously randomized to a coupon for discounted placebo soft-gel capsules by our collaborators, Vireo.
  Interventions: Other: Receipt of Coupon for Placebo Soft-Gel Capsule
- Coupon for a Discounted High THC Product (Other): We will observe participants who were previously randomized to a coupon for discounted 4.29 mg THC/0.72 mg CBD soft-gel capsules by our collaborators, Vireo.
  Interventions: Other: Receipt of Coupon for High THC Soft-Gel Capsule
- Coupon for a Discounted Equal THC and CBD Product (Other): We will observe participants who were previously randomized to a coupon for discounted 2.5 mg THC/2.5 mg CBD soft-gel capsules by our collaborators, Vireo.
  Interventions: Other: Receipt of Coupon for Equal THC and CBD Soft-Gel Capsule
- Coupon for a Discounted High CBD Product (Other): We will observe participants who were previously randomized to a coupon for discounted 0.25 mg THC/4.75 mg CBD soft-gel capsules by our collaborators, Vireo.
  Interventions: Other: Receipt of Coupon for High CBD Soft-Gel Capsule

INTERVENTIONS:
Other: Receipt of Coupon for Placebo Soft-Gel Capsule — The investigators will follow participants who were randomized to receive a coupon for placebo soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
  Placebo (0:0) Softgel, 0mg THC and 0mg CBD per cap, Bottle of 30 caps
  Arms: Coupon for a Discounted Placebo Product
Other: Receipt of Coupon for High THC Soft-Gel Capsule — The investigators will follow participants who were randomized to receive a coupon for high THC soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
  Vireo Yellow (6:1) Softgel, 4.29mg THC and 0.72mg CBD per cap, Bottle of 30 caps
  Arms: Coupon for a Discounted High THC Product
Other: Receipt of Coupon for Equal THC and CBD Soft-Gel Capsule — The investigators will follow participants who were randomized to receive a coupon for equal THC and CBD soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
  Vireo Green (1:1) Softgel, 2.5mg THC and 2.5mg CBD per cap, Bottle of 30 caps
  Arms: Coupon for a Discounted Equal THC and CBD Product
Other: Receipt of Coupon for High CBD Soft-Gel Capsule — The investigators will follow participants who were randomized to receive a coupon for high CBD soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
  Vireo Indigo (1:19) Softgel, 0.25mg THC and 4.75mg CBD per cap, Bottle of 30 caps
  Arms: Coupon for a Discounted High CBD Product

SUMMARY:
This study will examine how medical cannabis use affects neuropathic pain, inflammation and adverse events in people living with HIV (PLWH) with neuropathic pain. The investigators will observe how varying ratios of tetrahydrocannabinol (THC) and cannabidiol (CBD) in medical cannabis impact neuropathic pain, inflammation and adverse events.

DETAILED DESCRIPTION:
This study will examine how medical cannabis use affects neuropathic pain in PLWH with neuropathic pain. The investigators will enroll adults with HIV who have a) neuropathic pain, b) are actively certified for medical cannabis, and c) intend to have soft gel capsule products dispensed at Vireo (medical cannabis dispensary). The investigators will observe how pain and inflammation change in participants after they are randomized to receive high THC:low CBD product, an equal THC:CBD product, a low THC:high CBD product, or placebo by our collaborator in a separate study. Over 14 weeks, data sources will include questionnaires, blood samples, urine samples; medical, pharmacy, and Prescription Monitoring Program (PMP) records. The primary independent variable will be type of medical cannabis product dispensed at dispensary, and the primary outcome will be self-reported pain.

ELIGIBILITY:
Inclusion criteria:

->=18 years old

* Diagnosis of HIV
* Fluency in English
* Active certification for medical cannabis
* ICD-10 diagnosis code for neuropathic pain, OR Neuropathic pain in problem list of electronic medical record, OR Neuropathic pain per medical cannabis certification form, OR Neuropathic Pain Questionnaire-Short Form>0

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete 14 weeks of study visits
* Medical cannabis use within 14 days of enrollment, and no medical cannabis dispensed within 30 days of enrollment
* Unique pain symptoms (e.g., multiple sclerosis, rheumatoid arthritis)
* Terminal illness
* Current or prior psychotic disorder
* Unregulated cannabis use in the past 14 days; opioid or cocaine use in the past 30 days
* Dispensed opioids within 30 days
* Non-steroidal anti-inflammatory use within 7 days prior to enrollment
* Steroid use within the past 14 days with duration of therapy >=21 days
* COVID vaccination or booster within 14 days of screening
* Active or acute cardiac disease based on clinician chart review.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepika E Slawek, MD, MPH, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Health System, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Conference of State Legislatures. State Medical Marijuana Laws. Published 2020. Updated 11/6/2020.
- [Background] New York State Department of Health. Medical Use of Marijuana Under the Compassionate Care Act. In. Vol 22018.
- [Background] Russo E, Guy GW. A tale of two cannabinoids: the therapeutic rationale for combining tetrahydrocannabinol and cannabidiol. Med Hypotheses. 2006;66(2):234-46. doi: 10.1016/j.mehy.2005.08.026. Epub 2005 Oct 4. PMID 16209908
- [Background] Merlin JS, Cen L, Praestgaard A, Turner M, Obando A, Alpert C, Woolston S, Casarett D, Kostman J, Gross R, Frank I. Pain and physical and psychological symptoms in ambulatory HIV patients in the current treatment era. J Pain Symptom Manage. 2012 Mar;43(3):638-45. doi: 10.1016/j.jpainsymman.2011.04.019. Epub 2011 Nov 23. PMID 22115794
- [Background] Newshan G, Bennett J, Holman S. Pain and other symptoms in ambulatory HIV patients in the age of highly active antiretroviral therapy. J Assoc Nurses AIDS Care. 2002 Jul-Aug;13(4):78-83. doi: 10.1016/S1055-3290(06)60373-7. PMID 12149887
- [Background] Harding R, Lampe FC, Norwood S, Date HL, Clucas C, Fisher M, Johnson M, Edwards S, Anderson J, Sherr L. Symptoms are highly prevalent among HIV outpatients and associated with poor adherence and unprotected sexual intercourse. Sex Transm Infect. 2010 Dec;86(7):520-4. doi: 10.1136/sti.2009.038505. Epub 2010 Jun 15. PMID 20551235
- [Background] Silverberg MJ, Jacobson LP, French AL, Witt MD, Gange SJ. Age and racial/ethnic differences in the prevalence of reported symptoms in human immunodeficiency virus-infected persons on antiretroviral therapy. J Pain Symptom Manage. 2009 Aug;38(2):197-207. doi: 10.1016/j.jpainsymman.2008.08.007. Epub 2009 Mar 28. PMID 19329274
- [Background] Cervia LD, McGowan JP, Weseley AJ. Clinical and demographic variables related to pain in HIV-infected individuals treated with effective, combination antiretroviral therapy (cART). Pain Med. 2010 Apr;11(4):498-503. doi: 10.1111/j.1526-4637.2010.00802.x. Epub 2010 Mar 4. PMID 20210870
- [Background] Lee KA, Gay C, Portillo CJ, Coggins T, Davis H, Pullinger CR, Aouizerat BE. Symptom experience in HIV-infected adults: a function of demographic and clinical characteristics. J Pain Symptom Manage. 2009 Dec;38(6):882-93. doi: 10.1016/j.jpainsymman.2009.05.013. PMID 19811886
- [Background] Merlin JS, Westfall AO, Raper JL, Zinski A, Norton WE, Willig JH, Gross R, Ritchie CS, Saag MS, Mugavero MJ. Pain, mood, and substance abuse in HIV: implications for clinic visit utilization, antiretroviral therapy adherence, and virologic failure. J Acquir Immune Defic Syndr. 2012 Oct 1;61(2):164-70. doi: 10.1097/QAI.0b013e3182662215. PMID 22766967
- [Background] Miaskowski C, Penko JM, Guzman D, Mattson JE, Bangsberg DR, Kushel MB. Occurrence and characteristics of chronic pain in a community-based cohort of indigent adults living with HIV infection. J Pain. 2011 Sep;12(9):1004-16. doi: 10.1016/j.jpain.2011.04.002. PMID 21684218
- [Background] Bruce RD, Merlin J, Lum PJ, Ahmed E, Alexander C, Corbett AH, Foley K, Leonard K, Treisman GJ, Selwyn P. 2017 HIV Medicine Association of Infectious Diseases Society of America Clinical Practice Guideline for the Management of Chronic Pain in Patients Living With Human Immunodeficiency Virus. Clin Infect Dis. 2017 Oct 30;65(10):1601-1606. doi: 10.1093/cid/cix848. PMID 29091230
- [Background] Phillips TJC, Brown M, Ramirez JD, Perkins J, Woldeamanuel YW, Williams ACC, Orengo C, Bennett DLH, Bodi I, Cox S, Maier C, Krumova EK, Rice ASC. Sensory, psychological, and metabolic dysfunction in HIV-associated peripheral neuropathy: A cross-sectional deep profiling study. Pain. 2014 Sep;155(9):1846-1860. doi: 10.1016/j.pain.2014.06.014. Epub 2014 Jun 26. PMID 24973717
- [Background] Merlin JS. Chronic Pain in Patients With HIV Infection: What Clinicians Need To Know. Top Antivir Med. 2015 Aug-Sep;23(3):120-4. PMID 26518396
- [Background] Van der Watt JJ, Wilkinson KA, Wilkinson RJ, Heckmann JM. Plasma cytokine profiles in HIV-1 infected patients developing neuropathic symptoms shortly after commencing antiretroviral therapy: a case-control study. BMC Infect Dis. 2014 Feb 10;14:71. doi: 10.1186/1471-2334-14-71. PMID 24512313
- [Background] Manchikanti L, Cash KA, Damron KS, Manchukonda R, Pampati V, McManus CD. Controlled substance abuse and illicit drug use in chronic pain patients: An evaluation of multiple variables. Pain Physician. 2006 Jul;9(3):215-25. PMID 16886030
- [Background] Merlin JS, Zinski A, Norton WE, Ritchie CS, Saag MS, Mugavero MJ, Treisman G, Hooten WM. A conceptual framework for understanding chronic pain in patients with HIV. Pain Pract. 2014 Mar;14(3):207-16. doi: 10.1111/papr.12052. Epub 2013 Apr 1. PMID 23551857
- [Background] Bair MJ, Robinson RL, Katon W, Kroenke K. Depression and pain comorbidity: a literature review. Arch Intern Med. 2003 Nov 10;163(20):2433-45. doi: 10.1001/archinte.163.20.2433. PMID 14609780
- [Background] Fishbain DA. Approaches to treatment decisions for psychiatric comorbidity in the management of the chronic pain patient. Med Clin North Am. 1999 May;83(3):737-60, vii. doi: 10.1016/s0025-7125(05)70132-2. PMID 10386123
- [Background] Morasco BJ, Gritzner S, Lewis L, Oldham R, Turk DC, Dobscha SK. Systematic review of prevalence, correlates, and treatment outcomes for chronic non-cancer pain in patients with comorbid substance use disorder. Pain. 2011 Mar;152(3):488-497. doi: 10.1016/j.pain.2010.10.009. Epub 2010 Dec 23. PMID 21185119
- [Background] Rivera-Rivera Y, Garcia Y, Toro V, Cappas N, Lopez P, Yamamura Y, Rivera-Amill V. Depression Correlates with Increased Plasma Levels of Inflammatory Cytokines and a Dysregulated Oxidant/Antioxidant Balance in HIV-1-Infected Subjects Undergoing Antiretroviral Therapy. J Clin Cell Immunol. 2014 Dec;5(6):1000276. doi: 10.4172/2155-9899.1000276. PMID 25674354
- [Background] Surratt HL, Kurtz SP, Levi-Minzi MA, Cicero TJ, Tsuyuki K, O'Grady CL. Pain treatment and antiretroviral medication adherence among vulnerable HIV-positive patients. AIDS Patient Care STDS. 2015 Apr;29(4):186-92. doi: 10.1089/apc.2014.0104. Epub 2014 Jul 1. PMID 24984142
- [Background] Merlin JS, Long D, Becker WC, Cachay ER, Christopoulos KA, Claborn K, Crane HM, Edelman EJ, Harding R, Kertesz SG, Liebschutz JM, Mathews WC, Mugavero MJ, Napravnik S, C O'Cleirigh C, Saag MS, Starrels JL, Gross R. Brief Report: The Association of Chronic Pain and Long-Term Opioid Therapy With HIV Treatment Outcomes. J Acquir Immune Defic Syndr. 2018 Sep 1;79(1):77-82. doi: 10.1097/QAI.0000000000001741. PMID 29771793
- [Background] Abrams DI, Jay CA, Shade SB, Vizoso H, Reda H, Press S, Kelly ME, Rowbotham MC, Petersen KL. Cannabis in painful HIV-associated sensory neuropathy: a randomized placebo-controlled trial. Neurology. 2007 Feb 13;68(7):515-21. doi: 10.1212/01.wnl.0000253187.66183.9c. PMID 17296917
- [Background] Ellis RJ, Toperoff W, Vaida F, van den Brande G, Gonzales J, Gouaux B, Bentley H, Atkinson JH. Smoked medicinal cannabis for neuropathic pain in HIV: a randomized, crossover clinical trial. Neuropsychopharmacology. 2009 Feb;34(3):672-80. doi: 10.1038/npp.2008.120. Epub 2008 Aug 6. PMID 18688212
- [Background] Vergara D, Bidwell LC, Gaudino R, Torres A, Du G, Ruthenburg TC, deCesare K, Land DP, Hutchison KE, Kane NC. Compromised External Validity: Federally Produced Cannabis Does Not Reflect Legal Markets. Sci Rep. 2017 Apr 19;7:46528. doi: 10.1038/srep46528. PMID 28422145
- [Background] Volkow ND, Compton WM, Weiss SR. Adverse health effects of marijuana use. N Engl J Med. 2014 Aug 28;371(9):879. doi: 10.1056/NEJMc1407928. No abstract available. PMID 25162899
- [Background] Patton GC, Coffey C, Carlin JB, Degenhardt L, Lynskey M, Hall W. Cannabis use and mental health in young people: cohort study. BMJ. 2002 Nov 23;325(7374):1195-8. doi: 10.1136/bmj.325.7374.1195. PMID 12446533
- [Background] Caspi A, Moffitt TE, Cannon M, McClay J, Murray R, Harrington H, Taylor A, Arseneault L, Williams B, Braithwaite A, Poulton R, Craig IW. Moderation of the effect of adolescent-onset cannabis use on adult psychosis by a functional polymorphism in the catechol-O-methyltransferase gene: longitudinal evidence of a gene X environment interaction. Biol Psychiatry. 2005 May 15;57(10):1117-27. doi: 10.1016/j.biopsych.2005.01.026. PMID 15866551
- [Background] Bonn-Miller MO, Oser ML, Bucossi MM, Trafton JA. Cannabis use and HIV antiretroviral therapy adherence and HIV-related symptoms. J Behav Med. 2014 Feb;37(1):1-10. doi: 10.1007/s10865-012-9458-5. Epub 2012 Oct 7. PMID 23054178
- [Background] Slawson G, Milloy MJ, Balneaves L, Simo A, Guillemi S, Hogg R, Montaner J, Wood E, Kerr T. High-intensity cannabis use and adherence to antiretroviral therapy among people who use illicit drugs in a Canadian setting. AIDS Behav. 2015 Jan;19(1):120-7. doi: 10.1007/s10461-014-0847-3. PMID 25012624
- [Background] Keller S, Bann CM, Dodd SL, Schein J, Mendoza TR, Cleeland CS. Validity of the brief pain inventory for use in documenting the outcomes of patients with noncancer pain. Clin J Pain. 2004 Sep-Oct;20(5):309-18. doi: 10.1097/00002508-200409000-00005. PMID 15322437
- [Background] Moriarty AS, Gilbody S, McMillan D, Manea L. Screening and case finding for major depressive disorder using the Patient Health Questionnaire (PHQ-9): a meta-analysis. Gen Hosp Psychiatry. 2015 Nov-Dec;37(6):567-76. doi: 10.1016/j.genhosppsych.2015.06.012. Epub 2015 Jun 18. PMID 26195347
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] McLellan AT, Kushner H, Metzger D, Peters R, Smith I, Grissom G, Pettinati H, Argeriou M. The Fifth Edition of the Addiction Severity Index. J Subst Abuse Treat. 1992;9(3):199-213. doi: 10.1016/0740-5472(92)90062-s. PMID 1334156
- [Background] Greene B, Bernardo L, Thompson M, Loughead J, Ashare R. Behavioral Economic Strategies to Improve Enrollment Rates in Clinical Research: Embedded Recruitment Pilot Trial. JMIR Form Res. 2023 Jul 21;7:e47121. doi: 10.2196/47121. PMID 37477975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-five (35) participants were consented and enrolled into the study. One participant completed screening, consent and enrollment, but then did not want to be randomized into one of the coupon categories (study arms). As such, 34 patients were randomized into the study.
Groups:
- Coupon for a Discounted Placebo Product: Participants who were previously randomized to a coupon for discounted placebo soft-gel capsules by the collaborators, Vireo, will be observed.
  Receipt of Coupon for Placebo Soft-Gel Capsule: The investigators will follow participants who were randomized to receive a coupon for placebo soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
- Coupon for a Discounted High Tetrahydrocannabinol (THC) Product: Participants who were previously randomized to a coupon for discounted 4.3 mg tetrahydrocannabinol (THC)/0.7 mg cannabidiol (CBD) soft-gel capsules by the collaborators, Vireo, will be observed.
  Receipt of Coupon for High THC Soft-Gel Capsule: The investigators will follow participants who were randomized to receive a coupon for high THC soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
- Coupon for a Discounted Equal THC and Cannabidiol (CBD) Product: Participants who were previously randomized to a coupon for discounted 2.5 mg THC/2.5 mg CBD soft-gel capsules by the collaborators, Vireo, will be observed.
  Receipt of Coupon for Equal THC and CBD Soft-Gel Capsule: The investigators will follow participants who were randomized to receive a coupon for equal THC and CBD soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
- Coupon for a Discounted High CBD Product: Participants who were previously randomized to a coupon for discounted 0.2 mg THC/4.8 mg CBD soft-gel capsules by the collaborators, Vireo, will be observed.
  Receipt of Coupon for High CBD Soft-Gel Capsule: The investigators will follow participants who were randomized to receive a coupon for high CBD soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
Period: Overall Study
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High Tetrahydrocannabinol (THC) Product | Coupon for a Discounted Equal THC and Cannabidiol (CBD) Product | Coupon for a Discounted High CBD Product
Started | 9 | 8 | 9 | 8
Completed | 8 | 6 | 8 | 8
Not Completed | 1 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — No longer interested in participating | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Coupon for a Discounted High THC Product: Participants who were previously randomized to a coupon for discounted 4.3 mg THC/0.7 mg CBD soft-gel capsules by the collaborators, Vireo, will be observed.
  Receipt of Coupon for High THC Soft-Gel Capsule: The investigators will follow participants who were randomized to receive a coupon for high THC soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
- Coupon for a Discounted Equal THC and CBD Product: Participants who were previously randomized to a coupon for discounted 2.5 mg THC/2.5 mg CBD soft-gel capsules by the collaborators, Vireo, will be observed.
  Receipt of Coupon for Equal THC and CBD Soft-Gel Capsule: The investigators will follow participants who were randomized to receive a coupon for equal THC and CBD soft-gel capsule medical cannabis products by our collaborators at Vireo medical cannabis dispensary in a separate study
- Total: Total of all reporting groups
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product | Total
Number analyzed (Participants) | 9 | 8 | 9 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (10.9) | 52.5 (9.65) | 55.9 (10.7) | 61.8 (6.96) | 55.0 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 7 | 4 | 16
  Male | 9 | 3 | 2 | 4 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 6 | 4 | 17
  Not Hispanic or Latino | 3 | 7 | 3 | 4 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 5 | 4 | 18
  White | 3 | 1 | 0 | 1 | 5
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 9 | 8 | 34
CD4 Count [Mean (Standard Deviation); unit: cells/uL] — Blood samples were collected at baseline for CD4 counts. CD4 counts measure the number of CD4 T-lymphocytes, a type of white blood cell crucial for a healthy immune system and can serve as an indicator of HIV progression as well as how effectively HIV medications are working. For people with HIV infection, a CD4 count between 500-1500 cells/microliter is considered normal, and a count <200 cells/microliter signals advanced immune damage. Results are summarized by study arm and reported in cells/microliter (cells/uL). Population: Baseline CD4 count results were unable to be obtained from 1 participant in the High CBD arm and 1 participant in the Placebo arm.
  cells/uL
    number analyzed (Participants) | 8 | 8 | 9 | 7 | 32
    (all) | 658.63 (414.89) | 699.12 (185.88) | 828.78 (444.96) | 621.43 (458.37) | 708.47 (375.61)
Pain Severity Score [Mean (Standard Deviation); unit: score on a scale] — Pain Severity was measured at baseline using the Brief Pain Inventory (BPI) pain severity subscale. The BPI Pain Severity subscale uses a 0-10 numerical rating scale where 0 = "No pain at all" and 10 = "Pain as bad as you can imagine; completely interferes" such that higher scores were associated with increased Pain Severity. Participants were asked to assign a score to their pain, on average, over the prior week. Scores were summarized by study arm using basic descriptive statistics.
  score on a scale | 6.22 (2.54) | 7.63 (1.18) | 8.56 (1.13) | 7.5 (1.85) | 7.47 (1.68)
Circulating levels of Pro-Inflammatory and Anti-inflammatory Cytokines [Mean (Standard Deviation); unit: NPX value] — Circulating test levels of recent inflammation (based on a panel of inflammatory markers) was analyzed at baseline. Blood draws for circulating levels of pro-inflammatory (i.e., TNFa and IL-6) and anti-inflammatory (i.e., IL-10 and IL-6) cytokines were collected, processed, and analyzed using an O-link assay which uses normal protein expression (NPX) values expressed on a log2 scale, where a higher value indicates a higher protein level. Baseline results for each cytokine type are summarized by study arm using basic descriptive statistics. Population: Samples were not obtained from a number of participants at baseline and there were quality control issues with a couple of the sample. Accordingly, no baseline results data are available for these patients.
  NPX value
    Interleukin-10 (IL-10): number analyzed (Participants) | 5 | 7 | 8 | 6 | 26
    Interleukin-10 (IL-10) | 4.01 (0.53) | 3.7 (0.3) | 3.98 (0.68) | 3.69 (0.35) | 3.84 (0.47)
    Interleukin-4 (IL-4): number analyzed (Participants) | 5 | 7 | 8 | 6 | 26
    Interleukin-4 (IL-4) | 0.94 (0.77) | 0.47 (0.25) | 0.55 (0.49) | 0.81 (1.22) | 0.66 (0.65)
    Tumor Necrosis Factor Alpha (TNFa): number analyzed (Participants) | 5 | 7 | 8 | 6 | 26
    Tumor Necrosis Factor Alpha (TNFa) | 4.32 (0.89) | 3.95 (0.31) | 4.11 (0.49) | 3.97 (0.24) | 4.08 (0.46)
    Interleukin-6 (IL-6): number analyzed (Participants) | 5 | 7 | 8 | 6 | 26
    Interleukin-6 (IL-6) | 4.2 (0.73) | 4.17 (1.11) | 4.42 (0.67) | 4.52 (1.19) | 4.33 (0.92)
Antiretroviral Medication Adherence Score [Mean (Standard Deviation); unit: score on a scale] — Antiretroviral medication adherence was assessed at baseline using the Visual Analog Scale (VAS) of antiretroviral therapy (ART) adherence. This is an ordinal scale representing the percentage of medication taken to what had been administered. Participants were presented with a visual ranging from 0%-100% scaled at 10% increments and asked to provide a best guess as to how much medicine was taken over the past 30 days with 0% signifying no medication, 50% signifying half, and 100% signifying that all medication was taken. Scores are summarized by study arm using descriptive statistics. Population: A number of participants bypassed this question stating that they did not want to answer and skipped over it in the baseline questionnaire. No data from these participants was able to be collected/reported.
  score on a scale
    number analyzed (Participants) | 4 | 4 | 3 | 4 | 15
    (all) | 9.25 (1.5) | 10 (0) | 8 (3.46) | 8.25 (2.36) | 8.93 (1.72)
HIV Viral Load Suppression [Mean (Standard Deviation); unit: copies/mL] — HIV viral load was measured at baseline. Blood draws were obtained and samples were processed, analyzed, and quantified using the Abbott RealTime HIV-1 Viral Load assay. Results were summarized and HIV viral load values were reported in copies/milliliter (copies/mL). A high HIV viral load in the blood is associated with increased risk of disease progression and HIV transmission.
  copies/mL | 9560.33 (29836.6) | 0 (0) | 4.67 (13.2) | 18193.38 (5000.73) | 6812.71 (9078.06)
Depression Score [Mean (Standard Deviation); unit: score on a scale] — Depression score was measured at baseline using the Center for Epidemiologic Studies Depression (CES-D) questionnaire. The CES-D questionnaire is a 20-item screening tool used to assess the severity/frequency of depressive symptoms over the past week. Participants were asked to rate each of the 20 items on a 4-point Likert scale ranging from 0 ("Rarely/none of the time") to 3 ("Most/all of the time"), yielding an overall possible range of 0-60 (questions 4, 8, 12, and 16 were reverse-scored), such that higher scores indicated greater severity/frequency of depressive symptoms. Population: 4 participants did not complete the Depression questionnaire during baseline visit. No data from these participants was able to be collected/reported.
  score on a scale
    number analyzed (Participants) | 7 | 7 | 8 | 8 | 30
    (all) | 24.14 (11.61) | 23 (9.93) | 16.37 (7.93) | 17.88 (11.19) | 20.13 (10.12)
Anxiety Score [Mean (Standard Deviation); unit: score on a scale] — Anxiety score was measured at baseline using the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 is a 7-item screening tool used to assess the severity of anxiety-related symptoms. Participants were asked to rate each of the 7 items using a 4-point Likert scale ranging from 0 ("Not at all") to 3 ("Nearly every day") to indicate how long they have been bothered by the problems listed over the prior 2-week period, yielding an overall possible score of 0-21, with higher scores being indicative of worsening anxiety. Scores were summarized by study arm using basic descriptive statistics. Population: 4 participants did not complete the Anxiety questionnaire during baseline visit. No data from these participants was able to be collected/reported.
  score on a scale
    number analyzed (Participants) | 7 | 7 | 8 | 8 | 30
    (all) | 12.43 (6.85) | 5.71 (3.09) | 9.62 (6.14) | 7.38 (6.59) | 8.77 (5.71)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Severity Score
Description: Change in self-reported Pain Severity was measured at weekly intervals from baseline through 14 weeks using the Brief Pain Inventory (BPI) pain severity subscale. The BPI Pain Severity subscale uses a 0-10 numerical rating scale where 0 = "No pain at all" and 10 = "Pain as bad as you can imagine; completely interferes" such that higher scores were associated with increased Pain Severity. Participants were asked to assign a score to their pain, on average, over the prior week. Scores were summarized by study arm. For purposes of this study change in Pain Severity scores from baseline to 14 weeks following intervention were summarized and reported with positive values being indicative of increased pain severity compared to baseline and negative values being indicative of decreased pain severity compared to baseline.
Time Frame: At weekly intervals from Baseline to 14 weeks
Population: Number of participants analyzed is summarized for each arm/group at each week in the table below. Reasons for variability in the number of participants analyzed is attributable to missed virtual visits or incomplete data collection during specific timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
Number analyzed (Participants) | 9 | 8 | 9 | 8
score on a scale
  Week 1: number analyzed (Participants) | 9 | 7 | 7 | 8
  Week 1 | 6.44 (2.07) | 6.86 (2.27) | 8 (2.38) | 7.37 (2.5)
  Week 2: number analyzed (Participants) | 8 | 6 | 8 | 8
  Week 2 | 5.87 (3.09) | 6.67 (2.58) | 7.37 (1.76) | 6.75 (2.43)
  Week 3: number analyzed (Participants) | 9 | 8 | 7 | 8
  Week 3 | 5.22 (3.15) | 5.86 (2.23) | 7.57 (2.25) | 6.37 (2.92)
  Week 4: number analyzed (Participants) | 8 | 7 | 7 | 8
  Week 4 | 3.87 (2.64) | 6.28 (2.63) | 7.14 (2.73) | 6.375 (2.92)
  Week 5: number analyzed (Participants) | 9 | 5 | 7 | 6
  Week 5 | 4 (2.87) | 3 (2.34) | 7 (2.23) | 6.17 (2.71)
  Week 6: number analyzed (Participants) | 8 | 7 | 8 | 8
  Week 6 | 4.37 (2.72) | 5.14 (3.43) | 6.25 (2.37) | 5.37 (2.77)
  Week 7: number analyzed (Participants) | 9 | 7 | 8 | 8
  Week 7 | 4.11 (3.62) | 5.57 (2.29) | 6 (2.2) | 5.5 (3.07)
  Week 8: number analyzed (Participants) | 8 | 7 | 8 | 7
  Week 8 | 4.25 (3.11) | 4.86 (3.67) | 6 (2.56) | 6.57 (2.69)
  Week 9: number analyzed (Participants) | 9 | 6 | 7 | 7
  Week 9 | 3.44 (2.92) | 5.5 (4.63) | 5.28 (3.03) | 4.14 (2.97)
  Week 10: number analyzed (Participants) | 9 | 7 | 5 | 6
  Week 10 | 4.22 (3.73) | 5 (3.16) | 7.6 (2.07) | 5.33 (2.8)
  Week 11: number analyzed (Participants) | 9 | 8 | 6 | 8
  Week 11 | 3.88 (3.72) | 4.75 (2.96) | 6.83 (3.37) | 5.37 (2.97)
  Week 12: number analyzed (Participants) | 9 | 8 | 8 | 7
  Week 12 | 3.78 (3.67) | 6.37 (3.89) | 5.87 (3.18) | 6.14 (2.61)
  Week 13: number analyzed (Participants) | 9 | 8 | 7 | 8
  Week 13 | 3.55 (3.21) | 5 (3.21) | 5.43 (3.15) | 5.63 (2.5)
  Week 14: number analyzed (Participants) | 9 | 8 | 7 | 8
  Week 14 | -3 (2.39) | -2.625 (2.77) | -3.28 (2.36) | -1.88 (2.1)
Statistical Analysis 1: Comparison: Coupon for a Discounted High THC Product vs Coupon for a Discounted High CBD Product; The study team hypothesized that participants randomized to coupons for high THC products would have greater reduction in self-reported pain severity than high CBD, equal parts THC and CBD, or placebo; Test type: Superiority; p = 0.0303, Mixed Models Analysis — A mixed effects model was completed with Arm 2 as the reference; There were no adjustments for any covariates; Beta = -2.6185, 95% CI 2-sided [-4.98 to -0.25] — Arm 2 was the comparison arm
Statistical Analysis 2: Comparison: Coupon for a Discounted Placebo Product vs Coupon for a Discounted High THC Product; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4851, Mixed Models Analysis — A mixed effects model was completed with Arm 2 as the reference; There were no adjustments for any covariates; Beta = -0.8424 — Arm 2 was the comparison arm
Statistical Analysis 3: Comparison: Coupon for a Discounted High THC Product vs Coupon for a Discounted Equal THC and CBD Product; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6165, Mixed Models Analysis — A mixed effects model was completed with Arm 2 as the reference; There were no adjustments for any covariates; Beta = -0.6038 — Arm 2 was the comparison arm

2. Secondary Outcome: Change in Circulating Levels of Anti-inflammatory Cytokines - Interleukin-10 (IL-10)
Description: Change in circulating test levels of recent inflammation (based on a panel of inflammatory markers) from baseline to 14 weeks was analyzed. Blood draws for circulating levels of pro- and anti-inflammatory cytokines were collected, processed, and analyzed using an O-link assay which uses normal protein expression (NPX) values expressed on a log2 scale, where a higher value indicates a higher protein level. Results for IL-10 are summarized by study arm using basic descriptive statistics. For purposes of this study change in circulating levels of IL-10 from baseline to 14 weeks following intervention were summarized and reported. Samples were collected at two time points prior to the intervention and the results from these analyses were averaged and compared to the 14-week results.
Time Frame: From Baseline to 14 weeks
Population: Samples were not obtained from a number of participants at baseline and there were quality control issues with a couple of the samples. Accordingly, no change from baseline results data are available for these patients.
Measure: Mean (Standard Deviation); unit: NPX value
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
Number analyzed (Participants) | 5 | 7 | 8 | 6
NPX value | 0.15 (1.12) | 0.41 (0.83) | 0.11 (0.44) | 0.65 (0.85)
Statistical Analysis 1: Comparison: Coupon for a Discounted Placebo Product vs Coupon for a Discounted High THC Product vs Coupon for a Discounted Equal THC and CBD Product vs Coupon for a Discounted High CBD Product; The study team hypothesized that anti-inflammatory cytokines (IL-4 and IL-10) would have greater increase in participants randomized to coupons for high CBD products than the other arms; Test type: Superiority — An ANOVA test with mean change in NPX values was completed; p = 0.6, ANOVA; Three degrees of freedom (3 DoF); F value (F-test) = 0.63

3. Secondary Outcome: Change in Circulating Levels of Anti-inflammatory Cytokines - Interleukin-4 (IL-4)
Description: Change in circulating test levels of recent inflammation (based on a panel of inflammatory markers) from baseline to 14 weeks was analyzed. Blood draws for circulating levels of pro- and anti-inflammatory cytokines were collected, processed, and analyzed using an O-link assay which uses normal protein expression (NPX) values expressed on a log2 scale, where a higher value indicates a higher protein level. Results for IL-4 are summarized by study arm using basic descriptive statistics. For purposes of this study change in circulating levels of IL-4 from baseline to 14 weeks following intervention were summarized and reported. Samples were collected at two time points prior to the intervention and the results from these analyses were averaged and compared to the 14-week results.
Time Frame: From Baseline to 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: NPX value
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
Number analyzed (Participants) | 5 | 7 | 8 | 6
NPX value | -0.33 (0.57) | -0.21 (0.48) | 0.02 (0.5) | 0.07 (0.54)
Statistical Analysis 1: Comparison: Coupon for a Discounted Placebo Product vs Coupon for a Discounted High THC Product vs Coupon for a Discounted Equal THC and CBD Product vs Coupon for a Discounted High CBD Product; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — An ANOVA test with mean change in NPX values was completed; p = 0.49, ANOVA; Three degrees of freedom (3 DoF); F value (F-test) = 0.83

4. Secondary Outcome: Change in Circulating Levels of Pro-inflammatory Cytokines - Tumor Necrosis Factor Alpha (TNFa)
Description: Change in circulating test levels of recent inflammation (based on a panel of inflammatory markers) from baseline to 14 weeks was analyzed. Blood draws for circulating levels of pro- and anti-inflammatory cytokines were collected, processed, and analyzed using an O-link assay which uses normal protein expression (NPX) values expressed on a log2 scale, where a higher value indicates a higher protein level. Results for TNFa are summarized by study arm using basic descriptive statistics. For purposes of this study change in circulating levels of TNFa from baseline to 14 weeks following intervention were summarized and reported. Samples were collected at two time points prior to the intervention and the results from these analyses were averaged and compared to the 14-week results.
Time Frame: From Baseline to 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: NPX value
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
Number analyzed (Participants) | 5 | 7 | 8 | 6
NPX value | -0.02 (0.64) | 0.03 (0.37) | 0.05 (0.18) | -0.18 (0.24)
Statistical Analysis 1: Comparison: Coupon for a Discounted Placebo Product vs Coupon for a Discounted High THC Product vs Coupon for a Discounted Equal THC and CBD Product vs Coupon for a Discounted High CBD Product; The study team hypothesized that pro-inflammatory cytokines (TNFa and IL-6) would have greater reduction in participants randomized to coupons for high CBD products than the other arms; Test type: Superiority — An ANOVA test with mean change in NPX values was completed; p = 0.66, ANOVA; Three degrees of freedom (3 DoF); F value (F-test) = 0.53

5. Secondary Outcome: Change in Circulating Levels of Pro-inflammatory Cytokines - Interleukin-6 (IL-6)
Description: Change in circulating test levels of recent inflammation (based on a panel of inflammatory markers) from baseline to 14 weeks was analyzed. Blood draws for circulating levels of pro- and anti-inflammatory cytokines were collected, processed, and analyzed using an O-link assay which uses normal protein expression (NPX) values expressed on a log2 scale, where a higher value indicates a higher protein level. Results for IL-6 are summarized by study arm using basic descriptive statistics. For purposes of this study change in circulating levels of IL-6 from baseline to 14 weeks following intervention were summarized and reported. Samples were collected at two time points prior to the intervention and the results from these analyses were averaged and compared to the 14-week results.
Time Frame: From Baseline to 14 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: NPX value
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
Number analyzed (Participants) | 5 | 7 | 8 | 6
NPX value | 0.24 (0.73) | 0.11 (1.58) | -0.18 (0.83) | -0.09 (0.33)
Statistical Analysis 1: Comparison: Coupon for a Discounted Placebo Product vs Coupon for a Discounted High THC Product vs Coupon for a Discounted Equal THC and CBD Product vs Coupon for a Discounted High CBD Product; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — An ANOVA test with mean change in NPX values was completed; p = 0.88, ANOVA; Three degrees of freedom (3 DoF); F value (F-test) = 0.21

6. Secondary Outcome: Change in Antiretroviral Medication Adherence Score
Description: Change in Antiretroviral medication adherence from baseline to 14 weeks was assessed using the Visual Analog Scale (VAS) of antiretroviral therapy (ART) adherence. This is an ordinal scale representing the percentage of medication taken to that which had been administered. Participants were presented with a visual ranging from 0% to 100% scaled at 10% increments and asked to provide a best guess as to how much medicine was taken over the prior 30 days with 0% signifying no medication, 50% signifying half of administered medication taken, and 100% signifying that every single dose of medication was taken. Higher scores were indicative of increased medication adherence. Scores were summarized by study arm. For purposes of this study change in antiretroviral adherence score from baseline to 14 weeks following intervention was summarized and reported. Positive values are indicative of increased medication adherence from baseline and negative values are indicative of decreased adherence.
Time Frame: From Baseline to 14 weeks
Population: A number of participants bypassed this question stating that they did not want to answer and skipped over it in the baseline questionnaire. No change from baseline results data was able to be reported from these participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
Number analyzed (Participants) | 4 | 4 | 3 | 4
score on a scale | -1 (2.708) | 0 (0) | 2 (3.46) | 1 (2)
Statistical Analysis 1: Comparison: Coupon for a Discounted Placebo Product vs Coupon for a Discounted High THC Product vs Coupon for a Discounted Equal THC and CBD Product vs Coupon for a Discounted High CBD Product; The study team hypothesized that participants randomized to coupons for high THC products would have poorer Antiretroviral (ARV) medication adherence than those randomized to coupons for high CBD, equal parts THC and CBD, or placebo; Test type: Superiority — An ANOVA test with the mean change in adherence score was completed; p = 0.39, ANOVA; Three degrees of freedom (3 DoF); F value (F-test) = 1.11

7. Secondary Outcome: Change in HIV Viral Load Suppression
Description: Change in HIV viral load suppression from baseline was measured and assessed at 14 weeks. Blood draws were obtained at baseline and 14 weeks following intervention and samples were processed, analyzed, and quantified using the Abbott RealTime HIV-1 Viral Load assay. Results were summarized and HIV viral load values were reported in copies/milliliter (copies/mL). For purposes of this study change in HIV viral load from baseline to 14 weeks following intervention were summarized and reported. Positive values are indicative of increased HIV viral load levels compared to baseline and negative values are indicative of decreased/suppressed HIV viral load levels compared to baseline. A high HIV viral load in the blood is associated with increased risk of disease progression and HIV transmission.
Time Frame: From Baseline to 14 weeks
Population: Samples were unable to be obtained from several participants at baseline. No change from baseline results data was able to be reported from these participants.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
Number analyzed (Participants) | 7 | 7 | 8 | 7
copies/mL | -12270.43 (32267.19) | 7.7 (20.4) | -5 (14.9) | 3737 (9891.17)
Statistical Analysis 1: Comparison: Coupon for a Discounted Placebo Product vs Coupon for a Discounted High THC Product vs Coupon for a Discounted Equal THC and CBD Product vs Coupon for a Discounted High CBD Product; The study team hypothesized that participants randomized to coupons for high THC products would have less suppressed HIV viral load than those randomized to coupons for high CBD, equal parts THC and CBD or placebo; Test type: Superiority — An ANOVA test with mean change in HIV viral load was completed; p = 0.31, ANOVA; Three degrees of freedom (3 DoF); F value (F-test) = 1.25

8. Secondary Outcome: Change in Depression Score
Description: Change in Depression score was measured at baseline and 14 weeks using the Center for Epidemiologic Studies Depression (CES-D) questionnaire. The CES-D questionnaire is a 20-item screening tool used to assess the severity and frequency of depressive symptoms. Participants were asked to rate each of the 20 items using a 4-point Likert scale ranging from 0 ("Rarely/none of the time") to 3 ("Most/all of the time") to describe symptoms over the prior week (Questions, 4, 8, 12, and 16 were reverse-scored). Scores were summed to yield an overall possible scoring range of 0-60 with higher scores being indicative of increased severity/frequency of depressive symptoms. For purposes of this study change in depression score from baseline to 14 weeks following intervention was summarized. Positive values are indicative of increased depressive symptom severity/frequency compared to baseline and negative values are indicative of decreased depressive symptom severity/frequency compared to baseline.
Time Frame: From Baseline to 14 weeks
Population: 4 participants did not complete the Depression questionnaire during baseline visit. No change from baseline results data was able to be reported from these participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
Number analyzed (Participants) | 7 | 7 | 8 | 8
score on a scale | -9.71 (6.6) | -9 (9.39) | -3.56 (7.07) | -2.25 (5.52)
Statistical Analysis 1: Comparison: Coupon for a Discounted Placebo Product vs Coupon for a Discounted High THC Product vs Coupon for a Discounted Equal THC and CBD Product vs Coupon for a Discounted High CBD Product; The study team hypothesized that participants randomized to coupons for high THC products would have greater depression than those randomized to coupons for high CBD, equal parts THC and CBD, or placebo; Test type: Superiority — An ANOVA test with the mean change in depression score was completed; p = 0.13, ANOVA; Three degrees of freedom (3 DoF); F value (F-test) = 2.04

9. Secondary Outcome: Change in Anxiety Score
Description: Change in Anxiety score was measured and assessed at baseline and 14 weeks using the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 is a 7-item screening tool used to assess the severity of anxiety-related symptoms. Participants were asked to rate each of the 7 items using a 4-point Likert scale ranging from 0 ("Not at all") to 3 ("Nearly every day") to indicate how long they have been bothered by the problems listed over the prior 2-week period, yielding an overall possible score of 0-21, with higher scores being indicative of worsening anxiety. Scores were summarized by study arm. For purposes of this study change in anxiety score from baseline to 14 weeks following intervention was summarized and reported. Positive values are indicative of increased anxiety symptoms compared to baseline and negative values are indicative of decreased anxiety symptoms compared to baseline.
Time Frame: From Baseline to 14 weeks
Population: 4 participants did not complete the Anxiety questionnaire during baseline visit. No change from baseline results data was able to be reported from these participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
Number analyzed (Participants) | 7 | 7 | 8 | 8
score on a scale | -5.71 (4.07) | -1.43 (2.57) | -1.75 (4.68) | -1.12 (6.03)
Statistical Analysis 1: Comparison: Coupon for a Discounted Placebo Product vs Coupon for a Discounted High THC Product vs Coupon for a Discounted Equal THC and CBD Product vs Coupon for a Discounted High CBD Product; The study team hypothesized that participants randomized to coupons for high THC products would have greater anxiety than those randomized to coupons for high CBD, equal parts THC and CBD, or placebo; Test type: Superiority — An ANOVA test with the mean change in anxiety score was completed; p = 0.22, ANOVA; Three degrees of freedom (3 DoF); F value (F-test) = 1.58

ADVERSE EVENTS:
Time Frame: Up to approximately 14 weeks following intervention
Arm/Group | Coupon for a Discounted Placebo Product | Coupon for a Discounted High THC Product | Coupon for a Discounted Equal THC and CBD Product | Coupon for a Discounted High CBD Product
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/8 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 1/9 | 1/8 | 0/9 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coupon for a Discounted Placebo Product (N=9) | Coupon for a Discounted High THC Product (N=8) | Coupon for a Discounted Equal THC and CBD Product (N=9) | Coupon for a Discounted High CBD Product (N=8)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coupon for a Discounted Placebo Product (N=9) | Coupon for a Discounted High THC Product (N=8) | Coupon for a Discounted Equal THC and CBD Product (N=9) | Coupon for a Discounted High CBD Product (N=8)
Peripheral Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study did not reach its intended sample size as it was originally designed to enroll 100 participants. Accordingly, the study is underpowered and there may be limitations in the generalizability of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT05554146/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT05554146/ICF_001.pdf